CLINICAL TRIAL: NCT05548673
Title: Evaluatıon of the Effıcıency of Stress Management Traınıng Applıed to Nursıng Students (Happy Nursıng Student)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Kamile ÖNER, PhD, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Ankara Yildirim Beyazıt Univ
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stress
Keywords: Nursing education; Stress; Stress management education; Happy nursing student

STUDY DESIGN:
Intervention Model Description: It was conducted in a mixed method as a randomized controlled intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Stress management training was applied to the experimental group for eight weeks in sessions of 60-90 minutes once a week.
  Interventions: Behavioral: Psychoeducation
- Control group. (No Intervention): No action was taken on the students in the control group.

INTERVENTIONS:
Behavioral: Psychoeducation — The implementation phase is planned for Ankara Yıldırım Beyazıt University (AYBU) Nursing Faculty students. The stress management training program, which consists of eight sessions, is completed in 8 weeks, once a week.
  Arms: Experimental Group

SUMMARY:
This research was conducted to determine the effect of stress management education on the perceived stress levels, coping styles, self-esteem, happiness and general health of nursing students. It was conducted in a mixed method as a randomized controlled intervention study.

DETAILED DESCRIPTION:
The research was carried out at Ankara Yıldırım Beyazıt University in the 2021-2022 academic year. 20 nursing students were assigned to the experimental group and 20 to the control group. Stress management training was applied to the experimental group selected in the research for eight weeks in 60-90-minute sessions once a week. No action was taken on the students in the control group. Quantitative data, Socio-demographic data form, Perceived Stress Scale (PSS), Scale of Stress-Coping Styles (SCSS), Rosenberg Self-Esteem Scale (RSES), Oxford Happiness Scale-Short Form (OHQ-SF) and General Health Questionnaire-12 (GHQ-12). Qualitative data were collected through a semi-structured focus group interview form with the experimental group after the training. The analysis of the data was made using the IBM SPSS 25.0 statistical package program.

ELIGIBILITY:
Inclusion Criteria:

* Having completed the age of 18
* Being a registered (ongoing) Nursing Program student at Ankara Yıldırım Beyazıt University
* Having no problem attending school
* Being open to communication and cooperation
* Not having been diagnosed with any mental illness
* No diagnosis of mental illness in first degree relatives
* Not having a situation that would prevent them from participating in the trainings (Students will be included in the study after being evaluated within the scope of the SCL90-R test results).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Quantitative method - The Numerical Rating Scale(NRS) | five months
  It was applied to the experimental and control groups in order to quantitatively measure the effectiveness of stress management training, which was applied for 8 weeks.
Qualitative methot-Semi-structured focus group interview form | one weeks
  It was applied to evaluate the opinions and suggestions of the experimental group about the training program.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | five months
  The education given was used to determine the perceived stress levels of the students. While the scores obtained from the PSS range from 0 to 56, a high score from the scale indicates that the person is highly stressed.
Scale of Stress-Coping Styles (SCSS) | five months
  The training given was used to determine the students' levels of coping with stress. Higher scores indicate that the person uses that style more. The total score is a minimum of 30 and a maximum of 120 points.
Rosenberg Self-Esteem Scale (RSES) | five months
  The education given was used to determine the self-esteem levels of the students. Scale items score between 0 and 6, and self-esteem; are evaluated as high (0-1 points), medium (2-4 points) and low (5-6 points). In other words, the higher the score a person gets from the scale, the lower the self-esteem level is.
Oxford Happiness Scale-Short Form (OHQ-SF) | five months
  The education given was used to determine the happiness levels of the students. A score between 7 and 35 is taken from the scale. A high score from the scale indicates a high level of happiness.
General Health Questionnaire-12 (GHQ-12) | five months
  The education given was used to determine the general health levels of the students. The scale is likert style and consists of 4 options. The first two options are evaluated as "0" and the last two options as "1" points. The highest possible score is "12" and the lowest score is "0". Those who score 4 or more on the scale are evaluated as "high", those with 2-3 points as "medium", and those with less than 2 points as "low". The higher the score obtained from the scale, the higher the probability of psychiatric disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül ÖZKAN, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazit University, Ankara, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No